CLINICAL TRIAL: NCT00242177
Title: Pilot Test of ACTOS in Multiple Sclerosis: Safety and Tolerability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Douglas L Feinstein, Research Professor, Dept Anesthesiology, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-0547
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Relapsing, Remitting; Autoimmune disease
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Recurrence; Autoimmune Diseases | interventions — Pioglitazone

INTERVENTIONS:
Drug: ACTOS (Pioglitazone)

SUMMARY:
The purpose of this study is to determine whether an already FDA approved drug is safe and tolerable in Relapsing Remitting Multiple Sclerosis patients.

DETAILED DESCRIPTION:
1. Current treatments for Multiple Sclerosis (MS) only partially reduce the relapse rate or improve symptoms, have to be injected, and have side effects. In animal models of MS, the FDA-approved oral anti-diabetic drug ACTOS prevented and reduced symptoms. ACTOS has a good safety profile in diabetics and healthy volunteers, but it's effects in MS are not known. This trial will test the safety of taking daily ACTOS in Relapsing Remitting MS (RRMS) patients, the most common form of MS. Subjects will take ACTOS or a non active pill (placebo) every day, and during the trial the safety of the drug will be tested by doing blood tests for certain enzymes related to liver function, for glucose levels, by having the blood pressure measured, and having other routine laboratory blood tests carried out. The safety of ACTOS on MS disease will be tested by doing neurological examinations, Magnetic Resonance Imaging (MRI, a method which gives an image of the damage MS causes in brain), and other blood tests to make sure that the MS symptoms are not made worse by ACTOS. Findings that ACTOS is safe and tolerated in RRMS patients will help provide the basis for designing Phase II trials.
2. Subjects will be selected who have been diagnosed with RR-MS and who are taking the drug Avonex or Rebif to treat their MS symptoms. Subjects will be randomized to receive either ACTOS (30 mg) or a non-active tablet (placebo). Both the subjects and the investigator will be blinded meaning no-one will know which pill they are given. The subjects will take one pill daily by mouth for up to 18 months, the length of the trial. During the trial, subjects will be examined 8 times. At each visit about 3 tablespoons (30cc) of blood will be taken for tests. Subjects will have a total of 3 MRI scans done during the trial (at months 0, 5, and 12) to test if ACTOS effects the number or size of plaques in brain. At each visit the subjects will also have vital signs checked, and a urine pregnancy test performed
3. ACTOS can cause fluid retention which may cause or increase the risk of heart damage. ACTOS can cause mild weight gain or anemia (low hemoglobin levels). ACTOS can cause mild hypoglycemia (low blood sugar levels). ACTOS can increase ovulation and increase risk of pregnancy. Since ACTOS is structurally related to Troglitazone, which was associated with liver damage and rare cases of liver failure, patients treated with ACTOS are carefully monitored for changes in liver enzyme levels. In other studies with ACTOS, the most common side effects were upper respiratory tract infections, sinusitis, muscle pain, tooth disorder, sore throat, headache and gas. ACTOS may have other side effects, such as heartburn, diarrhea, constipation, dizziness, abdominal fullness, nausea, and loose stools.

   MRI is a FDA approved safe procedure. Possible risks include feelings of anxiety or claustrophobia, or disturbance by noise made during the procedure. A safe contrast agent (gadolinium) will be used for MRI. Injection and insertion of the needle may cause minor pain, bruising, and/or infection at the injection site. Gadolinium may cause brief discomfort, tingling, or warmth in the lips, or metallic taste in the mouth, tingling in the arm, nausea, or headache. Very rarely, there may be an allergic reaction. A standard questionnaire will be used to determine the safety for each patient before an MRI.

   Blood sample collection has risks of edema, swelling, or infection at the site of withdrawal.

   We will discuss all of the above in the consent form as outlined in the form with the candidates.
4. There are no known benefits from participating in this trial; however the knowledge gained may benefit others in the future.
5. This trial will recruit 30 RR MS patients. Approximately 10 male and 20 female patients will be recruited, with about equal numbers coming from the UIC and Rush. Patients can be between the ages of 18-64 yrs, and will be obtained from outpatient clinics. Consent process will follow standardized forms.

ELIGIBILITY:
Inclusion Criteria:

Informed consent must be signed and dated Clinically or laboratory definite RR MS Mild symptoms, with current EDSS between 1 and 6.5, and ambulatory Currently taking, and history (>= 1 year) of taking Avonex or Rebif No relapses in past 3 months Historical annual relapse rate of >=1.0 for the past 2 years Male or female, age 18 to 65 No history of liver disease, hypoglycemia, or cardiac related diseases Ability to carry out requirements for participation Not meeting any exclusion criteria

Exclusion Criteria:

Not meeting all inclusion criteria If female, pregnant, or intent to become pregnant or breast feed during trial Unable to give written consent Unable to carry out requirements of trial History of other neurological disease History of cardiovascular disease History of liver disease History of hypoglycemia History of high blood pressure HIV positive Exacerbation within 90 days of enrollment Intolerance to MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-10; Study Completion 2005-10

PRIMARY OUTCOMES:
MRI with GD enhancement at visit 2, 5, 8
Blood test (CBC, Liver enzymes)at each visit
EDSS at each visit
MSFC at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Douglas L Feinstein, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Pershadsingh HA, Heneka MT, Saini R, Amin NM, Broeske DJ, Feinstein DL. Effect of pioglitazone treatment in a patient with secondary multiple sclerosis. J Neuroinflammation. 2004 Apr 20;1(1):3. doi: 10.1186/1742-2094-1-3. PMID 15285799
- [Background] Schmidt S, Moric E, Schmidt M, Sastre M, Feinstein DL, Heneka MT. Anti-inflammatory and antiproliferative actions of PPAR-gamma agonists on T lymphocytes derived from MS patients. J Leukoc Biol. 2004 Mar;75(3):478-85. doi: 10.1189/jlb.0803402. Epub 2003 Dec 4. PMID 14657213
- [Background] Feinstein DL, Galea E, Gavrilyuk V, Brosnan CF, Whitacre CC, Dumitrescu-Ozimek L, Landreth GE, Pershadsingh HA, Weinberg G, Heneka MT. Peroxisome proliferator-activated receptor-gamma agonists prevent experimental autoimmune encephalomyelitis. Ann Neurol. 2002 Jun;51(6):694-702. doi: 10.1002/ana.10206. PMID 12112074